CLINICAL TRIAL: NCT03186794
Title: Pilot Study Characterizing Aerobic Exercise in Women With Systemic Lupus Erythematosus (Exercise SLE Pilot).
Brief Title: Aerobic Exercise in Women With Systemic Lupus Erythematosus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research activities were suspended due to the COVID-19 pandemic
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 170111; 17-CC-0111
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-03

CONDITIONS: Systemic Lupus Erythematosus; Lupus; Autoimmune Disease; Rheumatic Disease
Keywords: Rehabilitation; Fatigue
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Rheumatic Diseases; Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic exercise training (AET) (Experimental): Participants with systemic lupus erythematosus participated in a 12-week aerobic exercise training program. Exercise was performed on a treadmill, three times a week for 30 minutes at target training intensity of 70 - 80% of heart rate reserve [0.7 to 0.8 * (peak heart rate - resting heart rate) + resting heart rate]
  Interventions: Other: Treadmill exercise training

INTERVENTIONS:
Other: Treadmill exercise training — 30 minutes of continuous treadmill walking at a target intensity or use of an interval approach in which walking at the target will be sustained at smaller training interval durations of no shorter than 5 minutes followed by an active rest interval that is no longer than 1.5 times the training interval until the subject achieves a total exercise time of 30 minutes, excluding the rest intervals. Each session will last about 60 minutes but slightly longer if an interval approach is used.

SUMMARY:
Background:

As many as 1.5 million Americans are living with systemic lupus erythematosus (Lupus). Lupus makes people very tired. It also makes it hard for people to be physically active. Studies have shown that aerobic exercise training helps people with heart or lung illnesses be less tired and more active. Researchers want to use an exercise training program on people with Lupus to see if it has the same results.

Objectives:

To find out if aerobic exercise helps people with Lupus be less tired and more active.

Eligibility:

Women ages 21-80 who have Lupus and are not physically active.

Design:

Participants will be screened with a medical history and physical exam. They will have heart and lung tests, as well as blood and urine tests. They will also answer questions about their quality of life and take a test that measures lupus activity.

The study will last 14-16 weeks.

For the first two study visits, participants will do treadmill exercise tests and answer more quality of life questions. For these treadmill tests, participants will wear sensors, a mask, or a mouthpiece while they exercise.

Participants will then begin exercise training, 3 times a week for 12 weeks. At each of these visits, they will walk very fast for 30 minutes on a track or a treadmill. Each visit will last about 1 hour.

At the halfway point of the study, participants will repeat some of the screening tests. This visit will last about 3 hours.

At the end of the study, participants will repeat the screening tests. They will also repeat the treadmill exercise tests.

DETAILED DESCRIPTION:
We propose a single-arm exploratory study to characterize the responses and adaptations to aerobic exercise in women who have mild to moderate systemic lupus erythematosus (SLE) uncomplicated by organ damage that would limit participation. This is a pilot study to provide additional preliminary data to support a future U01 application. Persistent, excessive fatigue is among the three most debilitating symptoms of SLE and is cited by as many as 50% of patients as the single most debilitating symptom. We have observed, in women with mild SLE, significant relationships among deficits in work capacity and oxygen consumption obtained during treadmill exercise and patient reported measures of fatigue severity. Clinically significant functional aerobic impairment was present in these women, suggesting an underlying pathophysiological limitation that restricted cardiorespiratory capacity to well below that expected to occur as a result of normal deconditioning due to a sedentary lifestyle and lack of physical activity. We have also observed prolonged rest to steady state metabolic transition during even submaximal exercise in women with SLE . At peak exercise, muscle oxygenation deficiency was apparent despite normal increases in central circulatory oxygen delivery to the active muscles. Muscle tissue studies in other laboratories have implicated muscle basal lamina thickening as an oxygen diffusion barrier, which could possibly diminish the rate of tissue oxygen uptake and restrict cardiorespiratory capacity. Aerobic exercise training could improve cardiorespiratory capacity in women with SLE and with that improvement precipitate a reduction in their fatigability, particularly if that fatigability is mediated by impaired cardiorespiratory function.

Our research team is uniquely qualified to undertake this research and is one of the few teams possessing the experience and background necessary for contributing to this novel, understudied, yet critical field of rehabilitation research. For example, in addition to Dr. Keyser's studies on cardiorespiratory dysfunction in women with SLE, our team has studied the effects of an intense aerobic exercise-training program in individuals who have pulmonary hypertension (PH) or interstitial lung disease (ILD), two conditions associated with autoimmune diseases such as SLE. In fact, several of the subjects had SLE and the majority had autoimmune diseases of somewhat similar etiology. Our results demonstrated improved cardiorespiratory function and diminished fatigability in these patients, without serious adverse events, following a 10-week regimen of intense aerobic exercise training. Adherence to the protocol was over 90% in both subject subsets and there were no serious adverse events in either of these groups.

Subjects of the proposed research will be between 21 and 80 years of age and living within a reasonable travel distance from the greater Washington D.C. area. Subjects will be recruited from the NIH/National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) Intramural Research Program (IRP) Lupus Clinics. All tests and exercise training will be conducted at the NIH Clinical Center. There will be a single treatment condition consisting of 12-weeks of supervised treadmill walking, three times a week, for 30 minutes per session, at an intensity of 70-80% of the subject's heart rate reserve.

The primary outcome measure for our trial will be the time taken to attain the anaerobic threshold, which is a performance marker of fatigability that is unaffected by patient motivation or perception. Secondary outcome variables will include other measures of cardiorespiratory capacity measured during a cardiopulmonary exercise test (CPET) with accompanying pulmonary gas exchange, central circulatory function (including heart function and an optional measures of peripheral blood flow), and muscle oxygenation analyses. A number of questionnaires will also be completed including: Fatigue Severity Scale, Patient Reported Outcomes Measurement Information System (PROMIS). All of these data will be obtained before and after aerobic exercise training.

Study Impact: Aerobic exercise is generally safe, inexpensive, and can easily be made available and accessible to almost everyone. It requires no approval by regulatory agencies and is thus available as a medically prescribed and supervised intervention almost immediately following confirmation of its safety and efficacy. Effective use of aerobic exercise training as a cardiorespiratory, rehabilitative intervention could have a high degree of impact on personal and public health outcomes.

ELIGIBILITY:
INCLUSION CRITERIA:

* Fulfilling 4 of the 11 American College of Rheumatology Criteria for the Classification of Systemic Lupus Erythematosus
* Age 21 to 80
* Female Gender
* BMI less than 40
* No primary or secondary medical conditions that would limit aerobic capacity or make exercise participation unsafe. (These conditions are found under the exclusion criteria listed below and include cardiovascular disease and cardiomyopathy, pulmonary and pulmonary vascular disease, stroke, significant hepatic or renal dysfunction, most cancers, diabetes mellitus, HIV infection, and peripheral vascular disease.)
* SELENA-SLEDAI score less than or equal to 4, maintained for at least three months. (C3 and C4 levels are measured as markers for stability and included in the SELENA-SLEDAI score if abnormal).
* No increase in doses of immunosuppressive medications (hydroxychloroquine, mycophenolate mofetil, azathioprine, methotrexate) for at least three months at the time of screening.
* No increase in the dose of prednisone or equivalent steroid in the past 3 months at the time of screening.
* Physically inactive, not participating in aerobic exercise training at heart rate above 60% maximum heart rate, 20 min/session or more, 2 or more days per week, within the last 6 months at the time of screening.
* Fatigue Severity Scale (FSS) composite score greater than or equal to 3 indicating the presence of clinically significant fatigue
* Subjects must be able to walk on a treadmill

EXCLUSION CRITERIA:

* Prednisone greater than or equal to 15 mg daily (or equivalent)
* Have started azathioprine, mycophenolate mofetil, methotrexate, cyclophosphamide or biologics within 3 months
* Rituximab infusion within 6 months
* Present symptoms of ischemic heart disease, right- or left-sided heart failure, cor pulmonale or pulmonary hypertension, dilated or hypertrophic cardiomyopathy or non- idiopathic cardiomyopathy
* Significant pulmonary dysfunction (obstructive, restrictive, or infectious pulmonary disease)
* Significant hepatic (LFT > 2 times of upper limit of normal) or renal dysfunction (GFR<45 ml/min)
* Deep vein thrombosis
* Chronic anticoagulation (with the exception of low dose aspirin) or a history of a bleeding disorder
* History or presence of any form of cancer other than skin cancer or cervical in-situ cancer
* History of cerebrovascular accident
* Orthopedic conditions that would limit performance of treadmill exercise tests or treadmill exercise training
* Current smoker or active substance abuse
* HIV infection
* Any medication that limit exercise capacity or the ability to adapt to aerobic exercise training (e.g. beta-blockers, anti-retroviral therapy for the treatment of HIV infection)
* Diabetes Mellitus
* Fibromyalgia: Determined at pre-screening visit, as per 2010 American College of Rheumatology (ACR) criteria for diagnosis of fibromyalgia
* Uncontrolled or untreated thyroid dysfunction: Determined by abnormal Thyroid Stimulating Hormone (TSH) level checked at the time of screening or within 3 months before screening visit.
* Currently pregnant, nursing or plan to become pregnant during the duration of the study
* Anemia (hemoglobin < 9 g/dl)
* Significant peripheral vascular disease
* Severe Raynaud's phenomenon
* Individuals unable to give informed consent

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited, de-identified samples may be available to other NIH intramural researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of results.
Access Criteria: Permission of PI and approval from the IRB prior to any research use of stored de-identified samples beyond the scope of this study.

REFERENCES:
- [Background] Keyser RE, Rus V, Cade WT, Kalappa N, Flores RH, Handwerger BS. Evidence for aerobic insufficiency in women with systemic Lupus erythematosus. Arthritis Rheum. 2003 Feb 15;49(1):16-22. doi: 10.1002/art.10926. PMID 12579589
- [Background] Keyser RE, Rus V, Mikdashi JA, Handwerger BS. Exploratory study on oxygen consumption on-kinetics during treadmill walking in women with systemic lupus erythematosus. Arch Phys Med Rehabil. 2010 Sep;91(9):1402-9. doi: 10.1016/j.apmr.2010.06.003. PMID 20801259
- [Background] Carvalho MR, Sato EI, Tebexreni AS, Heidecher RT, Schenkman S, Neto TL. Effects of supervised cardiovascular training program on exercise tolerance, aerobic capacity, and quality of life in patients with systemic lupus erythematosus. Arthritis Rheum. 2005 Dec 15;53(6):838-44. doi: 10.1002/art.21605. PMID 16342102
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-CC-0111.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 subjects were consented. 20 subjects started the study. 2 subjects were screen failure and 2 subjects were withdrawn due to pandemic closure.
Groups:
- Aerobic Exercise Training (AET): Participants with systemic lupus erythematosus participated in a 12-week aerobic exercise training program. Exercise was performed on a treadmill, three times a week for 30 minutes at target training intensity of 70 - 80% of heart rate reserve [(0.7 to 0.8 * peak heart rate - resting heart rate)+ resting heart rate]
Period: Overall Study
Arm/Group | Aerobic Exercise Training (AET)
Started | 20
Completed | 16
Not Completed | 4
Not completed — Physician Decision | 2
Not completed — Withdrawal due to COVID-19 pandemic closure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in the Time Taken to Attain the Anaerobic Threshold (AT)
Description: The anaerobic threshold (AT) is an objective measure of fatigability, and is determined from gas exchange variables during a cardiopulmonary exercise test (CPET). The effect of exercise training was examined by the change in the time taken to attain the AT by measuring the post-exercise training value minus the pre-exercise training value. A positive value indicates improvement in fatigability and a negative value indicates no improvement or worsening in fatigability. CPET measurement was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-cardiopulmonary exercise testing (CPET)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
Seconds | 93.3 (82.2)

2. Primary Outcome: Change in the Time Constant for Oxygen Uptake Kinetics
Description: The oxygen uptake kinetics is an objective measure of fatigability, determined from oxygen uptake measures during a square-wave exercise test. The time constant is the time taken to reach 63% of the steady state response. The effect of exercise training was examined by the change in the time constant by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in fatigability and a positive value indicates no improvement or worsening in fatigability. The square-wave exercise test was done before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-square-wave exercise test
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
Seconds | -12.6 (20.4)

3. Primary Outcome: Change in Performance Fatigability Index (PerfFI)
Description: The performance fatigability index (PerfFI) is a measure of fatigability. The PerfFI was determined during a 10-minute walk test (10MWT). The average velocity of 10MWT was divided by the average velocity achieved over the first 2.5 minutes (decline in performance), then further divided by the total distance walked on the 10MWT (an index of intensity) multiplied by 1000. The effect of exercise training was examined by the change in the PerfFI by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in fatigability and a positive value indicates no improvement or worsening in fatigability. The 10MWT measurement was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-10 minute walk test (10MWT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
Units on a scale | -0.12 (0.09)

4. Primary Outcome: Change in Perceived Fatigability Index (PercFI)
Description: The perceived fatigability index (PercFI) is a measure of fatigability. The PercFI was determined during a 10-minute walk test (10MWT) by rating their perceive tiredness on a 7-point Likert scale after the test. The score is divided by the total distance walked on the 10MWT, multiplied by 1000. The effect of exercise training was examined by the change in the PerfFI by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in fatigability and a positive value indicates no improvement or worsening in fatigability. The 10MWT measurement was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-10 minute walk test (10MWT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
Units on a scale | -0.43 (1.55)

5. Secondary Outcome: Change in Muscle Oxygenation
Description: Muscle oxygenation is indicated by tissue saturation index (TSI), which is the amount of oxygenated hemoglobin divided by total hemoglobin in percent. This is evaluated using near-infrared spectroscopy (NIRS) during the cardiopulmonary exercise test (CPET). Peak TSI is determined at the end of the CPET representing the lowest muscle oxygenation during volitional exercise. The effect of exercise training was examined by the change in peak TSI by measuring the post-exercise training value minus the pre-exercise training value. A negative value may indicate better muscle oxygenation capacity and a positive value may indicate no change or reduction in muscle oxygenation capacity. The CPET was performed before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who performed pre- and post-NIRS measurements during the cardiopulmonary exercise testing (CPET)
Measure: Mean (Standard Deviation); unit: Percentage of TSI signal
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
Percentage of TSI signal | -2.2 (2.8)

6. Secondary Outcome: Change in Cardiac Function
Description: Cardiac function is indicated by cardiac output, which is the amount of blood the heart pumps in 1 minute. It is defined mathematically as the product of the heart rate and cardiac stroke volume. This is measured using bioimpedance cardiography (a non-invasive method of capturing cardiodynamic variables) during the cardiopulmonary exercise test (CPET). Peak cardiac output is determined at the end of the CPET representing the highest cardiac output during volitional exercise. The effect of exercise training was examined by the change in peak cardiac output by measuring the post-exercise training value minus the pre-exercise training value. A positive value indicates improvement in cardiac function and a negative value indicates no change or worsening in cardiac function. The CPET was performed before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post bioimpedance cardiography measurements with CPET
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
L/min | 1.3 (4.1)

7. Secondary Outcome: Change in Fatigue Severity Scale (FSS)
Description: The Fatigue Severity Scale (FSS) is a 9-item questionnaire that assesses fatigue severity on a 7-point Likert scale. The FSS score is an average of the total score for the 9-items, with a minimum of 1 and a maximum of 7. A higher FSS score indicate more fatigue severity. The effect of exercise training was examined by the change in FSS average scores by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in fatigue severity and a positive value indicates no improvement or worsening in fatigue severity. The FSS questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-Fatigue Severity Scale (FSS) questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
score on a scale | -1.4 (1.0)

8. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Anxiety Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The anxiety domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more anxiety being measured. The effect of exercise training was examined by the change in anxiety domain by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in anxiety and a positive value indicates no improvement or worsening in anxiety. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | -3.5 (7.0)

9. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Depression Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The depression domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more depression being measured. The effect of exercise training was examined by the change in depression domain by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in depression and a positive value indicates no improvement or worsening in depression. The PROMIS-57 profile was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | -4.8 (6.4)

10. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Fatigue Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The fatigue domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate greater fatigue. The effect of exercise training was examined by the change in fatigue domain by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in fatigue and a positive value indicates no improvement or worsening in fatigue. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | -6.0 (4.5)

11. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Physical Function Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The Physical Function domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more physical function being measured. The effect of exercise training was examined by the change in physical function domain by measuring the post-exercise training value minus the pre-exercise training value. A positive value indicates improvement in physical function and a negative value indicates no improvement or worsening in physical function. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | 3.6 (4.8)

12. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Sleep Disturbance Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The Sleep Disturbance domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more sleep disturbance being measured. The effect of exercise training was examined by the change in sleep disturbance domain by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in sleep disturbance and a positive value indicates no improvement or worsening in sleep disturbance. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | -2.4 (4.3)

13. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Ability to Participate in Social Roles and Activities Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The ability to participate in social roles and activities domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more ability to participate in social roles and activities. The effect of exercise training was examined by the change in ability to participate in social roles and activities domain by measuring the post-exercise training value minus the pre-exercise training value. A positive value indicates improvement in ability to participate in social roles and activities and a negative value indicates no improvement or worsening in ability to participate in social roles and activities. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | 1.0 (5.3)

14. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Pain Interference Domain
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. The pain interference domain is scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. Higher scores indicate more pain interference being measured. The effect of exercise training was examined by the change in pain interference domain by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in pain interference and a positive value indicates no improvement or worsening in pain interference. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
T-score | -3.9 (10.8)

15. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS-57 Profile): Pain Intensity Score
Description: The PROMIS-57 profile is a self-reported questionnaire assessing quality of life in various domains. Pain intensity is scored from 0 to 10, with higher scores indicating greater pain intensity. The effect of exercise training was examined by the change in pain intensity domain by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in pain intensity and a positive value indicates no improvement or worsening in pain intensity. The PROMIS-57 profile questionnaire was done once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who completed pre- and post-PROMIS-57 profile questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
score on a scale | -0.9 (1.8)

16. Secondary Outcome: Change in Safety of Estrogen in Lupus Erythematosus, National Assessment Modification of Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI)
Description: SELENA-SLEDAI is a 24-item weighted index measure of disease activity at time of assessment or in the preceding 10 days. It consists of clinical and laboratory variables, with a minimum score of 0 and maximum score of 105. Higher scores represent greater disease activity. The effect of exercise training was examined by the change in SELENA-SLEDAI by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates improvement in disease activity and a positive value indicates no improvement or worsening in disease activity. The SELENA-SLEDAI was assessed once before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who were assessed for SELENA-SLEDAI at pre- and post-exercise program
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
score on a scale | -0.2 (1.0)

17. Secondary Outcome: Change in Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SLICC/ACR-DI)
Description: SLICC/ACR-DI is a 41-item instrument used to assess damage since lupus disease onset. Clinical assessment is made in 12 different organ systems, and a sum total from all organ scales are computed. A minimum score of 0 and a maximum score of 47 is possible with higher scores indicating more damage. The effect of exercise training was examined by the change in SLICC/ACR-DI by measuring the post-exercise training value minus the pre-exercise training value. A negative value indicates no change in damage since disease onset and a positive value indicates increase in damage since disease onset. The SLICC/ACR-DI was assessed before the start of the 12-week exercise program (pre) and repeated at the end of the 12-week exercise program (post).
Time Frame: Before 12-week intervention (Pre) and after 12-week intervention (Post)
Population: The analyses included only those subjects who were assessed for SLICC/ACR-DI at pre- and post-exercise program
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise Training (AET)
Number analyzed (Participants) | 16
score on a scale | 0.1 (0.3)

ADVERSE EVENTS:
Time Frame: 23 weeks
Arm/Group | Aerobic Exercise Training (AET)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Training (AET) (N=20)
Palpitations (Cardiac disorders) | 1
Presyncope (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Dermatitis allergic (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Oral pain (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03186794/Prot_SAP_000.pdf